CLINICAL TRIAL: NCT04631003
Title: Pilot Study for a Dynamic Testing for Intraoperative Diagnosis of Scapholunate Instability in Patients With a Concurrent Distal, Intra Articular Radius Fracture - A Prospective Clinical Trial
Brief Title: Intraoperativ Testing of Scapholunate Instability in Radius Fracture
Acronym: ScaLu
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spital Davos AG (Network)
Collaborators: AO Research Institute Davos (Other)
Responsible Party: Principal Investigator, Dr. Michael Villiger, Co-Director of Davos Sports & Health, Spital Davos AG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-02146
Record Dates: First submitted 2020-10-21; First posted 2020-11-16 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Radius; Dislocation Distal; Scapholunate Dissociation
Keywords: Scapholunary Instability; Distal, intra-articulare Radius Fracture; Dynamic Functional Testing; Arthro-CT; Scapholunate Dissociation; Scapholunate Advanced Collapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dynamic testing (Other): There are only one arm in this study. All patients get the same diagnostics and therapy. The preoperative assessments consist of an arthroCT of the wrist as well as the collection of demographic data, accident mechanism, medication intake, etc. within the scope of the usual medical history on the emergency ward. With the arthro-CT, in addition to the fracture balance, the proof of a possible rupture of the scapholunary tape apparatus takes place.
  The dynamic determination of the scapholunary instability takes place during the osteosynthesis of the radius fracture.
  With the dynamic functional test, the change of the scapholunary distance is assessed by illumination by movement of the wrist from the radial abduction into the ulnar abduction, before and after the execution of the osteosynthesis of the distal radius fracture.
  Subsequently, the results of the scapholunary dissociation of the arthro-CT are checked with the results of the intraoperative dynamic test for correlation.
  Interventions: Diagnostic Test: dynamic functional testing

INTERVENTIONS:
Diagnostic Test: dynamic functional testing — First, with an arthroCT of the wrist by intraarticular injection of contrast agent, a possible scaphulonary band lesion is detected. The surgeon does not yet know the findings of the possible ligament injury at this time, but he can assess the fracture in the CT. Subsequently, a dynamic functional test of the scapholunary distance is carried out intraoperatively under investigation with the modified Watson test before and after performing the osteosynthesis. For this purpose, the wrist is intraoperatively brought under pull on the thumb from a radial abduction into an ulnarabduction. In the presence of a scapholunary instability, a change in the distance of the scapholunary joint gap is shown here under illumination. Now the surgeon receives the finding of the Arthro-CT regarding an existing ligament injury. If necessary, this is treated in the same anaesthetic with a band seam and ossary transfixation.

SUMMARY:
Ligamental side injuries in distal radius fractures are not uncommon, but diagnosis is often difficult. Diagnosis with the simultaneous presence of a fracture is not very reliable and usually highly subjective.

5-64% of radius fractures are accompanied by injuries of the scapholunary ligament (SL). Intra-articular radius fractures have a significantly higher prevalence for SL dissociation, due to a greater energy transfer to the hand roots. In 5-10% of cases, distal, intra-articular radius fractures are associated with complete ruptures of the dorsal scapholunary band. The number of untreated SL band lesions in distal radius fractures is largely unknown.

If left untreated, scapholunary ligament lesions, with the simultaneous presence of a rupture of the dorsal ligament, (DIC) can lead to symptomatic carpal instability, therefore the correct diagnosis and adequate therapy is necessary even in the presence of a distal radius fracture.

Through the band ruptures, both the Os lunatum and the Os scaphoideum experience irregular motion. This leads to Dorsal Intercalated Segment Instability (DISI) and is reflected by the flexion of the os scaphoideum and the extension of the os lunatum radiologically in the lateral uptake with an increase of the scapholunary angle > 60° (usually maximum 45)° and the radioscaphoidal angle >15°.

An incorrect use can lead to the development of SLAC-wrist (Scapho-Lunate Advanced Collapse) over years, this risk should be reduced if possibel by recognizing the original injury.

With regard to this problem, we would like to establish a radiological, dynamic functional test, allowing scapholunary ligament lesions in distal radius fractures to be diagnosed intraoperatively.

DETAILED DESCRIPTION:
Radius fractures are the most common fractures in adulthood and account for approximately 17.5% of all fractures. The most common distal radius fractures are approximately 57-66% extra-articular (AO type A), followed by completely articular fractures (AO type C) with 25-35% and the least rare partial articular fractures (AO type B) with 9-15%.

The fracture mechanism of distal radius fractures is in most cases a fall on the extended wrist, less often a high-energy trauma. It is not uncommon for there to be additional accompanying ligamental injuries, which are easily overlooked.

5-64% of intraarticular radius fractures are accompanied by injuries of the scapholunary ligament. However, most of these studies are carried out in smaller series, with only one exception. A scapholunary band lesion can occur in isolation or in combination with a distal radius fracture, scaphoid fracture or perilunary luxation. The prevalence of this ligament injury has not yet been sufficiently studied. Acute scapholunary ligament damage accompanying injury to a distal radius fracture, clinical testing of instability by means of the Watson provocation test is not possible due to pain. Thus, scapholunary dissociation is often initially overlooked. Additional later examinations by means of MRI or arthroscopy are necessary to diagnose the missed ligamentary injuries.

In 5-10% of cases, intraarticular radius fractures are associated with complete ruptures of the dorsal scapholunary band, which leads to symptomatic carpal instability with the simultaneous presence of a rupture of the dorsal ligamentum intercarpale (DIC). The number of untreated SL band lesions in distal radius fractures is largely unknown.

A scapholunary band lesion can be represented in different degrees of severity, depending on the still preserved portion of the scapholunary ligament and the surrounding extrinsical ligaments. Partial ruptures only lead to pain during movement and result in a slight restriction of scaphoid mobility. A scapholunary complete rupture, on the other hand, leads to a dissociation of ossa scaphoideum and lunatum, resulting in a Dorsal Intercalated Segment Instability (DISI). DISI malposition in turn leads in the long run to wrist osteoarthritis, called SLAC Wrist, with secondary development of osteoarthritis. The development of the full disease takes 10-20 years. The development of a SLAC Wrist can be counteracted preventively in which a scapholunary instability - also within the framework of a radius fracture - is detected at an early stage and correctly stabilized. However, the clinical relevance and the recommended treatment of scapholunary band rupture has not yet been definitively clarified.

A complete rupture of the scapholunary band alone does not necessarily lead to instability. Among other things, one study shows that the dorsal ligamentum intercaraple plays a very important role in the stabilization of the Os lunatum and the Os scaphoideum. Only with additional rupture of the ligamentum intercaraple dorsal, next to the ligamentum scapholunare, is there a Dorsal Intercalated Segment Instability.

The Os lunatum and the Os scaphoideum are coupled with each other by the scapholunary tape apparatus. With a complete rupture of the scapholunary band, both the os lunatum and the osscaphoideum follow the respective self-movement. The Os scaphoideum can no longer exert a force on the Os lunatum. Thus, without counter-action, there is a pulling force on the Os lunatum by the still intact ligamentum lunotriquetrale and da the Os lunatum palmar is wider than dorsal, the Os lunatum is pushed over time into a permanent position of the extension and palmaren dislocation. The Os scaphoideum, on the other hand, is anatomically "slanted" to the wrist axis and thus has a tendency towards flexion. The flexion of the Os scaphoideum leads to a dorsal subluxation of the os saphoideum to the fossa radialis. This phenomenone in turn leads to the Dorsal Intercalated Segment Instability (DISI). This is reflected by the flexion of the os scaphoideum and the extension of the os lunatum radiologically in the lateral uptake with an increase of the scapholunary angle > 60° (usually maximum 45)° and the radioscaphoidal angle >15° again. In the long run, this misalignment develops a wrist osteoarthritis called SLAC Wrist (Scapho-Lunate Advanced Collaps) with secondary development of osteoarthritis.

The effect of untreated scapholunary dissociation on wrist function is unknown despite abundant studies, but all with small series. However, it has been proven that they lead to symptomatic carpal instability, especially with additional rupture of the dorsal ligamentum intercarpale.

In a large study with 839 subjects, 25.6% of patients with distal radius fracture have scapholunary dissociation immediately after trauma, and only 13.4% continued to have a persi-sedate scpaholunary dissociation after repositioning and osteosynthesis. This can best be explained by stabilization due to the ligamentotaxis of the extrinsic carpal ligaments.

Another study showed an excellent long-term outcome in patients who were stable after volar plate osteosynthesis in distal radius fracture without surgical treatment of scapholunal dissociation in the functional test. Whereas a plaster cast leads to a worse outcome.

The Watson test, as used in clinical practice, is a provocation maneuver to diagnose a possible scapholic ligament lesion. Here, the Tubercel scaphoideum is fixed with the thumb and at the same time a wrist deviation from the radial duction and flexion into the ulnar duction and extension is performed. In the case of higher degree of instability in the sense of a complete rupture of the scapholunary band, the Watson test is positive if, in addition to pain, there is a palpable snap, due to a subluxation of the proximal scaphoid pole over dorsal radius at radial deviation and subsequent spontar position in the Fossa radii at Ulnadeviation. However, this test is not feasible with fresh radius fracture.

Accompanying scapholunary lesions in radius fractures are often underdiagnosed, although they are up to 54% in dislocated, distal radius fractures. A study shows that intraarticular radius fractures are twice more commonly associated with scapholic lesions than seen in radiological diagnostics, although there are conventional-radiological suggestive evidence for static scapholunary band lesions. It has been described that 60% of all scapholunary lesions show no abnormalities in conventional X-ray image and are therefore easily overlooked. A widened joint gap between Os scaphoideum and Os lunatum with a distance > 3mm as well as a tilting of the two carpalia to each other indicates apossible bandrupture but is not diagnostic. However, in patients with a distal radius fracture, more than half of patients with an SL distance > 3mm in ct also have an extension on the opposite side 38-52%. There are no uniform conventional-radiological criteria for determining the instability of the wrist and the scapholunary distance.

If none of the above abnormalities can be found in the conventional radiological images, however, a clinical suspicion of scpholunary dissociation leads to a MR tomography and an arthroscopy of the wrist. A computed tomography is not a sensitive modality for a band lesion. An arthro-CT, on the other hand, detects a ligament injury and is equivalent to arthro MRI with a sensitivity of 95%.

In current literature, the gold standard in the diagnosis of scapholunary ligament injuries is arthroscopy. Using wrist arthroscopy as an examination technique for scapholic ligamentions, 7-64% of all patients with a distal radius fracture show a rupture, in extra-articular radius fractures the incidence is lower with 7-33%. We do not require an indicative arthroscopy due to the increased risk of surgery and therefore also the risk of infection.

So far, there have been no studies that have used a clinical, dynamic functional test intraoperatively under screening, to assess scapholunary instability in intra-articular radius fractures. With intraoperative detection of an SL band lesion, this can be supplied surgically under the same anaesthesia with different methods such as a band seam, ossary reinsertion, carpal transfixing or combinations.

The core of the study is the actual intervention to which the patients commit themselves. In this case, patients receive a computed tomography of the affected wrist in distal, intra-articular radius fractures in order to preoperatively, in addition to fracture, diagnose possible concomitant ligamentic injuries, in particular of the scapholunary band rupture. Computed tomography without intraarticular contrast agent administration, on the other hand, is a standard for displaying the exact fracture curves in intraarticular, distal radius fractures.

Subsequently, the scpaholunary stability is checked under intraoperative investigation before and after osteosynthesis with a dynamic test modified by us. With the help of this test, a relevant, i.e. an unstable scpaholunary band lesion, is also to be diagnosed.

The aim of this study is to investigate scapholunous instability in distal, intraarticular radius fracture and thus to diagnose an accompanying scapholunary band rupture.

* Determination of the prevalence of scapholunary band lesions in distal, intraarticular radius fractures
* Detection of scapholic instability in distanceric, intraarticular radius fracture, with the intraoperative conduct of a modified, dynamic functional test under illumination

With the results, the intraoperative test will be able to be used in the future for the diagnosis of scapholunary band lesions and the detection of persistent carpal instability after osteosynthesis of radius fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a distal radius fracture that reaches into the wrist joint
* Age >16 and <80 years
* Signed informed consent
* Carrying out surgery of the radius fracture at Hospital of Davos

Exclusion Criteria:

* Age <16 and >80 years
* Contraindications for computer tomography or contrast agents
* Undislocated distal radius fractures that do not need meet criteria of stabilization with a plate (surgery)
* Serious illness that does not allow surgery
* Pregnancy
* Use of strong blood-thinning medications
* Severe coagulation disorder

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Dynamic Functional Testing | Through study completion, an average of 1 year
  Change in the distance between Os scaphoideum and Os lunatum in the dynamic function test under illumination in distal, intraarticular radius fracture and thus evidence of scapholunal instability. Intraoperatively, the scapholunary instability is investigated by means of a provocation test under illumination with the image converter. For this purpose, the wrist is moved from a radial abduction to an ulnarabduction under tension on the thumb in the ap recording. In the presence of a scapholunary dissociation, in the sense of an unstable band rupture, an increase in the scapholunary distance is shown.
  The obtained statement regarding a scapholunary dissociation by the function test must be verified with an arthro-CT.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Villiger, Principal Investigator — Spital Davos
Locations (1):
- Spital Davos AG, Davos Platz, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chim H, Moran SL. Wrist essentials: the diagnosis and management of scapholunate ligament injuries. Plast Reconstr Surg. 2014 Aug;134(2):312e-322e. doi: 10.1097/PRS.0000000000000423. PMID 25068352
- [Background] Forward DP, Lindau TR, Melsom DS. Intercarpal ligament injuries associated with fractures of the distal part of the radius. J Bone Joint Surg Am. 2007 Nov;89(11):2334-40. doi: 10.2106/JBJS.F.01537. PMID 17974874
- [Background] Geissler WB, Freeland AE, Savoie FH, McIntyre LW, Whipple TL. Intracarpal soft-tissue lesions associated with an intra-articular fracture of the distal end of the radius. J Bone Joint Surg Am. 1996 Mar;78(3):357-65. doi: 10.2106/00004623-199603000-00006. PMID 8613442
- [Background] Gunal I, Ozaksoy D, Altay T, Satoglu IS, Kazimoglu C, Sener M. Scapholunate dissociation associated with distal radius fractures. Eur J Orthop Surg Traumatol. 2013 Dec;23(8):877-81. doi: 10.1007/s00590-012-1093-x. Epub 2012 Oct 16. PMID 23412224
- [Background] Kitay A, Wolfe SW. Scapholunate instability: current concepts in diagnosis and management. J Hand Surg Am. 2012 Oct;37(10):2175-96. doi: 10.1016/j.jhsa.2012.07.035. PMID 23021178
- [Background] Lindau T, Arner M, Hagberg L. Intraarticular lesions in distal fractures of the radius in young adults. A descriptive arthroscopic study in 50 patients. J Hand Surg Br. 1997 Oct;22(5):638-43. doi: 10.1016/s0266-7681(97)80364-6. PMID 9752922
- [Background] Mitsuyasu H, Patterson RM, Shah MA, Buford WL, Iwamoto Y, Viegas SF. The role of the dorsal intercarpal ligament in dynamic and static scapholunate instability. J Hand Surg Am. 2004 Mar;29(2):279-88. doi: 10.1016/j.jhsa.2003.11.004. PMID 15043902
- [Background] Mrkonjic A, Lindau T, Geijer M, Tagil M. Arthroscopically diagnosed scapholunate ligament injuries associated with distal radial fractures: a 13- to 15-year follow-up. J Hand Surg Am. 2015 Jun;40(6):1077-82. doi: 10.1016/j.jhsa.2015.03.017. Epub 2015 Apr 30. PMID 25936737
- [Background] Pilny J, Kubes J, Hoza P, Mechl M, Visna P. [Scapholunate instability of the wrist following distal radius fracture]. Acta Chir Orthop Traumatol Cech. 2007 Feb;74(1):55-8. Czech. PMID 17331455
- [Background] Prommersberger KJ, Muhldorfer-Fodor M, Kalb K, Schmitt R, van Schoonhoven J. [Scapholunate lesions]. Unfallchirurg. 2014 Aug;117(8):723-37; quiz 738-9. doi: 10.1007/s00113-014-2621-4. German. PMID 25116013
- [Background] Richards RS, Bennett JD, Roth JH, Milne K Jr. Arthroscopic diagnosis of intra-articular soft tissue injuries associated with distal radial fractures. J Hand Surg Am. 1997 Sep;22(5):772-6. doi: 10.1016/S0363-5023(97)80068-8. PMID 9330132
- [Background] Short WH, Werner FW, Green JK, Masaoka S. Biomechanical evaluation of the ligamentous stabilizers of the scaphoid and lunate: Part II. J Hand Surg Am. 2005 Jan;30(1):24-34. doi: 10.1016/j.jhsa.2004.09.015. PMID 15680552
- [Background] Sun GTW, MacLean SBM, Alexander JJ, Woodman R, Bain GI. Association of scapholunate dissociation and two-part articular fractures of the distal radius. J Hand Surg Eur Vol. 2019 Jun;44(5):468-474. doi: 10.1177/1753193419826490. Epub 2019 Feb 6. PMID 30727814
- [Background] Suzuki D, Ono H, Furuta K, Katayama T, Akahane M, Omokawa S, Tanaka Y. Comparison of scapholunate distance measurements on plain radiography and computed tomography for the diagnosis of scapholunate instability associated with distal radius fracture. J Orthop Sci. 2014 May;19(3):465-70. doi: 10.1007/s00776-014-0533-3. Epub 2014 Jan 29. PMID 24473829
- [Background] Tang JB, Shi D, Gu YQ, Zhang QG. Can cast immobilization successfully treat scapholunate dissociation associated with distal radius fractures? J Hand Surg Am. 1996 Jul;21(4):583-90. doi: 10.1016/S0363-5023(96)80007-4. PMID 8842947